CLINICAL TRIAL: NCT06047262
Title: A Multi-Centre, Randomised, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of the Oral NLRP3 Inhibitor Dapansutrile in Subjects With Type 2 Diabetes Mellitus
Brief Title: Dapansutrile in Diabetes and Diabetes-Related Complications - Dapan-Dia
Acronym: Dapan-Dia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: European Union (Horizon Europe Programme) (Unknown); State Secretariat for Education Research and Innovation, Switzerland (Other); Olatec Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-01387; kt23Donath
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapansutrile

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 1000 mg dapansutrile (2 × 500mg tablets) administered twice a day from day 1 through the week 26 visit, inclusive. All tablets will be self-administered by mouth with water, with or without food.
  Interventions: Drug: Dapansutrile
- Control Group (Placebo Comparator): Matching placebo (2 tablets) administered twice a day from day 1 through the Week 26 visit, inclusive. All tablets will be self-administered by mouth with water, with or without food.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapansutrile — Patients receive investigational product.
  Other Names: 3-methanesulfonyl-propionitrile; OLT1177
  Arms: Intervention Group
Drug: Placebo — Patients receive placebo.
  Arms: Control Group

SUMMARY:
The aim of the study is to determine whether NLRP3 inhibition with dapansutrile represents a new pharmacological option for diabetes management with potential as an anti-inflammatory agent to also address micro- and macro-vascular risk and complications from diabetes.

DETAILED DESCRIPTION:
To date, no other oral NLRP3 inhibitor has sufficiently advanced in development to be tested in a chronic low-grade inflammatory disease such as type 2 diabetes mellitus over a period of 3 to 4 months as proposed in this trial. Based on the publicly available information, dapansutrile is the most advanced oral NLRP3 inhibitor in development. The rationale is built upon dapansutrile's clinical and extensive preclinical and safety findings, and from data in chronic animal toxicology studies to date, which together enable and support its investigation in select chronic low-grade inflammatory diseases. Therefore, the investigators have selected type 2 diabetes mellitus and its complications, including risk for cardiovascular disease, as a disease with clinical features of low-grade inflammation to further investigate the therapeutic potential of NLRP3 inhibition with dapansutrile.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2, Diabetes mellitus as defined by the criteria of the American Diabetes Association (ADA) Expert Committee on the Diagnosis and Classification of Diabetes Mellitus (see Appendix 1) and recognized by the World Health Organization (WHO, 2019), for at least 3 months prior to the Baseline Visit/Day 1
* HbA1c value of ≥ 7.7% to ≤ 11.0% at the Screening Visit.
* High-sensitivity C-reactive protein (hsCRP) ≥ 1.5 mg/L at the Screening Visit.
* Body mass index (BMI) ≥18 to ≤ 40 kg/m2 at the Screening Visit
* Acceptable overall medical condition to safely participate in the study and complete all study procedures (particularly with regard to cardiovascular, renal, and hepatic conditions), in the opinion of the Investigator

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus
* HbA1c value of ≤ 7.5% or ≥ 10.5% at the Baseline Visit/Day 1, as determined at point of care (local laboratory)
* Use of thiazolidinediones (glitazones), pramlintide, or short-acting insulin/insulin analogues (as bolus or premixed insulin) within 12 weeks prior to the Screening Visit
* Less than 80% compliance in taking investigational medicinal product by pill count during the Run-In Period, as assessed at the Baseline Visit/Day 1
* Significant weight loss (> 5 kg) in the 12 weeks prior to the Screening Visit
* Systolic blood pressure (BP) ≥ 160 mmHg, diastolic BP ≥ 100 mmHg, or resting heart rate (HR) ≥ 100 beats/minute at the Screening Visit
* Previous myocardial infarction, any cardiac surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c in blood of patients for dapansutrile compared to placebo | two time assessment at baseline and week 26
  Comparison of change in HbA1c for dapansutrile and placebo

SECONDARY OUTCOMES:
Change in HbA1c in blood of patients for dapansutrile compared to placebo | six time assessment at baseline and week 4, 8, 12, 16, 20
  Comparison of change in HbA1c for dapansutrile and placebo
Change in fasting plasma glucose for dapansutrile compared to placebo | seven time assessement at baseline and week 4, 8, 12, 16, 20, 26
  Comparison of change in fasting plasma glucose for dapansutrile and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y. Donath, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland